CLINICAL TRIAL: NCT05779839
Title: Fostering Caregiver Connections Via Intentional Technology Pairing for Caregivers of Patients With Alzheimer's Disease and Other Types of Dementia-Phase 2
Brief Title: A Study of Caregiver Connections Via Technology in Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Julie A. Fields, Ph.D., L.P., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-008835; R44AG065088 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-03-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Stress; Dementia; Alzheimer Disease; Lewy Body Dementia; Parkinson Disease Dementia; Frontotemporal Dementia
MeSH Terms: conditions — Caregiver Burden; Dementia; Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia | interventions — Algorithms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two different arms of the study: one where the algorithm matches individuals and one where matches are randomly assigned.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Algorithmically Matched (Experimental): Individuals that identify as a current and/or former caregiver for a person with dementia will be matched to other caregivers using an algorithm that matches a caregiver to another caregiver based on specific preferences each caregiver identifies in a questionnaire.
  Interventions: Behavioral: Algorithm
- Randomly Matched (Active Comparator): Individuals that identify as a current and/or former caregiver for a person with dementia will be randomly matched to other caregivers not based on the preferences they identified in a questionnaire.
  Interventions: Behavioral: Random Match

INTERVENTIONS:
Behavioral: Algorithm — For purpose of finding peer-to-peer support, current and/or former caregivers of persons with dementia will be matched using an algorithm. They can then choose make a connection and maintain a connection for the duration of the study.
  Arms: Algorithmically Matched
Behavioral: Random Match — For purpose of finding peer-to-peer support, current and/or former caregivers of persons with dementia will be randomly matched. They can then choose make a connection and maintain a connection for the duration of the study.
  Arms: Randomly Matched

SUMMARY:
This research is being done to develop a unique matching process for caregivers of persons living with dementia, such as Alzheimer's disease, Lewy body dementia, frontotemporal degeneration, or other dementia syndromes. Dementia caregivers often assume greater caregiving burden than do non-dementia caregivers, and the caregiving duration tends to be longer. Many caregivers do not have the adequate support they need. Peer-to-peer support has been shown to improve quality of life, more engagement with services, improve caregiver health, and reduce hospitalizations in the person they are caring for. This study will help determine whether caregivers of persons with dementia would find a technology-based caregiver matching program valuable for the purpose of emotional support.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have a family member that has been diagnosed with one of the following forms of dementia: Parkinson's/Lewy body dementia, any frontotemporal lobar degeneration dementia, or Alzheimer's dementia.
* The participant must identify as a care partner or caregiver who has contact with their loved one with dementia, in person or by phone, and provides social/emotional support and full or partial assistance with daily activities at least 3 days per week.
* The participant must have been caring for their loved one with dementia for at least 3 months.
* All participants must have access to a computer and be able to use the internet.
* All participants must be English speaking.
* All participants must agree to participate in the 15-month study, which includes completing questionnaires, brief "virtual" interactions with the study coordinator quarterly, and actively interacting with the website and potential matches.
* All participants must agree to follow-up contact throughout the duration of the study, which is anticipated to last 3 years.

Exclusion Criteria:

* Caregiver's loved one does not have a confirmed diagnosis of dementia.
* Caregiver is unable to provide consent.
* Caregiver was or has been in that role for less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Match Satisfaction Questionnaire | 12 months
  All participants will complete a match satisfaction questionnaire to assess whether being matched to a supportive caregiver via an algorithm based on personal preferences results in greater match satisfaction than being matched at random. Questions are scored from 0 to 4 with a possible total of 28.
  Scores are interpreted such that an overall total of: 0 - 7 = low satisfaction; 8-14 = medium/average satisfaction; 15-28 = high satisfaction
Change over time from Baseline Resilience to 12 months | Baseline, 12 months
  All participants will complete questions surveying resilience to determine whether caregivers randomized to algorithmic matching based on personal preferences will report a greater sense of resiliency after being matched than caregivers who are randomly matched.
Change over time from Baseline Quality of Life to 12 months | Baseline, 12 months
  All participants will complete questions surveying quality of life to determine whether caregivers randomized to algorithmic matching based on personal preferences will report improved quality of life after being matched than caregivers who are randomly matched.
Scale of Perceived Social Support | 12 months
  All participants will complete survey questions regarding perceived level of social support to assess impact on match satisfaction.

SECONDARY OUTCOMES:
Survey of Executive Skills | 12 months
  All participants will complete questions regarding executive functioning (e.g., flexibility, problem-solving) to determine whether the level of these skills relates to ease or difficulty in finding a satisfactory supportive caregiver match.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fields, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials